CLINICAL TRIAL: NCT05825313
Title: The Effect of Podcast Use in Nursing Education on Students' Speech Skill, Affective Awareness Towards Instruction and Success: A Randomized Controlled Trial
Brief Title: The Effect of Podcast Use Student's Skills in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hacer Ozel, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23.12.2021/4
Record Dates: First submitted 2023-03-03; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Podcast Group (Experimental): Podcast was applied to the experimental group.
  Interventions: Behavioral: Podcast Using
- Control Group (No Intervention): No intervention was applied to the control group.No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Podcast Using — Students in the experimental group listened to podcast episodes any time they desired following the course every week during the semester from February 2021 to June 2021.
  Arms: Podcast Group

SUMMARY:
This study was conducted to find out the effect of the use of podcasts in nursing education on nursing students' speaking skills, affective awareness towards instruction, and success in the course and to serve as a source for prospective studies on the topic.

DETAILED DESCRIPTION:
Objectives This study was conducted to find out the effect of the use of podcasts in nursing education on nursing students' speaking skills, affective awareness towards instruction, and success in the course and to serve as a source for prospective studies on the topic.

Design Randomized controlled trial. Settings A nursing faculty Participants Fourth-year nursing students who were studying at the faculty of nursing and were taking the "Academic Presentation Techniques" were randomly assigned to the experimental group (n=20) and the control group (n=20).

Methods Every week during the semester, students in the experimental group could listen to podcast episodes any time they desired following the course. Both before the podcast intervention and at the end of the semester, the Effective Speech Scale and the Scale of Affective Awareness Towards Instruction were administered to experimental and control groups. Final examination grades were evaluated as the indicator of success in the course.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old,
* Volunteer to participate in research

Exclusion Criteria:

* be under 18 years old,
* not voluntarily to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Speech Skills | Four months
  The student's speech skills were measured by Effective Speech Scale

SECONDARY OUTCOMES:
Affective Awareness Towards Instruction | Four months
  The student's affective awareness towards instruction were measured by affective awareness towards instruction understanding Affective Awareness Towards Instruction Scale.

OTHER OUTCOMES:
Success | Four months
  Course success is to complete the course with a successful grade. Final Exam form (questions) evaluated as a success criterion.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor S, Daly CS, MacArthur J, Borglin G, Booth RG. Podcasting in nursing and midwifery education: An integrative review. Nurse Educ Pract. 2020 Aug;47:102827. doi: 10.1016/j.nepr.2020.102827. Epub 2020 Jul 6. PMID 32763834